CLINICAL TRIAL: NCT06655064
Title: Prospective Observational Multicenter Registry Study to Assess the Impact & Long-Term Outcomes of 68Ga-PSMA-11 PET/CT Imaging Evaluations for Patients With Prostate Cancer (Newly Diagnosed, Suspected Recurrence P or Are Candidates for Radioligand Therapy)
Brief Title: Registry to Evaluate Long-Term Outcomes in Patients Who Undergo 68-Ga-PSMA-11 PET/CT Imaging Evaluations
Status: Terminated | Type: Observational
Why Stopped: Sponsor request
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Specialty Networks Research. (Network)
Responsible Party: Sponsor
Other Study IDs: 68Ga-PtableSMA-11-404
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: PSMA; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Newly Diagnosed: Patients who have been newly diagnosed with prostate cancer and have not received any prior treatment for prostate cancer and have undergone a 68Ga-PSMA-11 PET/CT imaging evaluation to evaluate potential spread of the disease.
  Interventions: Other: None- Observational
- Group 2: Previously Treated: Patients who have received previous treatment for prostate cancer and have and have undergone 68Ga-PSMA-11PET/CT imaging evaluation for suspected recurrence (demonstrated by elevated PSA levels).
  Interventions: Other: None- Observational
- Group 3: RLT Candidates: Patients who have metastatic prostate cancer and undergone a 68Ga-PSMA-11 PET/CT imaging evaluation for the initiation of RLT.
  Interventions: Other: None- Observational

INTERVENTIONS:
Other: None- Observational — None- Observational

SUMMARY:
The purpose of this observational research registry is to understand the real-world use of Illuccix PET/CT in prostate cancer, and how results from this testing impact patient's treatment and prostate cancer journey over time. It will follow subjects and the diagnostic testing and therapy they receive for their prostate cancer.

Subjects will not be administered any medical diagnostic testing or therapy that they would not have normally undergone outside of participation in the registry.

ELIGIBILITY:
Inclusion Criteria:

Participants will qualify for inclusion into Cohort 1, 2, or 3 only if they meet all the following criteria.

1. Be a biological male at birth who is ≥ 21 years of age at the time of informed consent.
2. Have undergone a 68Ga-PSMA-11 (Illuccix or Gozellix) PET/CT imaging evaluation within 60 days before enrolling in the study. (Prior imaging with alternate radioactive imaging agents are allowed, but enrollment imaging must be with 68Ga-PSMA-11(Illuccix or Gozellix).
3. Have histopathologically confirmed prostate adenocarcinoma.
4. Have a life expectancy of ≥ 6 months as determined by the investigator.
5. Participants intended for enrollment in Cohort 1: Patients who have been newly diagnosed with prostate cancer and have not received any prior treatment for prostate cancer and have undergone a 68Ga-PSMA-11 PET/CT imaging evaluation to evaluate potential spread of the disease.
6. Participants intended for enrollment in Cohort 2: Patients who have received previous treatment for prostate cancer and have and have undergone 68Ga-PSMA-11 PET/CT imaging evaluation for suspected recurrence (demonstrated by elevated PSA levels). Participants intended for enrollment in Cohort 3: Patients who have metastatic prostate cancer and undergone a 68Ga-PSMA-11 PET/CT imaging evaluation for the initiation of RLT.
7. Be willing and able to provide informed consent and comply with the protocol requirements.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply. All participants must NOT:

1. Have any medical condition or other circumstances that, in the opinion of the Investigator, compromises the safety of the participant, the ability of the participant to comply with protocol requirements, the ability of the participant to complete the study, or confound study outcomes by being unable to produce reliable data over the course of the study.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 500 participants will be enrolled at up to 15 investigative sites in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Prostate Cancer Long Term Outcomes | 3 years
  Long term outcomes of patients with newly diagnosed or recurrent disease prostate cancer or those being evaluated for radioligand therapy, who undergo 68Ga-PSMA-11PET/CT imaging for clinical management.

SECONDARY OUTCOMES:
Utilization of 68Ga-PSMA-1 PET/CT Imaging for Early Prostate Cancer Recurrence Detection | 1.5 years
  Utilization of 68Ga-PSMA-1 PET/CT imaging for early recurrence detection in patients with low PSA (< 0.2 ng/mL).
Patient Demographic and Clinical Characteristics | 1.5 years
  Demographic and clinical characteristics at time of imaging for prostate cancer patients undergoing 68Ga-PSMA-11 PET/CT imaging.
Utilization of 68Ga-PSMA-11 PET/CT Imaging for Initial Staging of Prostate Cancer | 1.5 years
  Utilization of 68Ga-PSMA-11 PET/CT imaging for initial staging in low risk to favorable intermediate risk [(Grade Group 1 and 2: Gleason score 6 and 7 (3+4)] prostate cancer patients.
Clinical Impact on Prostate Cancer Staging and Radioligand Treatment Planning | 1.5 years
  Clinical impact of 68Ga-PSMA-11PET/CT imaging on staging and treatment planning in prostate cancer patients considered for radioligand therapy.
Differential Use across Racial and Ethnic Groups | 3 years
  Differential use of 68Ga-PSMA-11 PET/CT imaging across racial and ethnic groups.
Conventional Imaging | 3 years
  Utilization of 68Ga-PSMA-11PET/CT imaging in initial evaluation vs repeat conventional imaging in treatment planning decisions for patients with new and recurrent prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Aimal Ahmed, MD, Study Director — Telix Pharmaceuticals
Locations (9):
- United States (9):
  - Valley Urology, Fresno, California
  - Urology Associates of Central California, Fresno, California
  - Urological Associates of Western Colorado, Grand Junction, Colorado
  - Idaho Urologic Institute, Meridian, Idaho
  - Comprehensive Urology, Royal Oak, Michigan
  - Urology Nevada, Reno, Nevada
  - Oregon Urologic Institute, Springfield, Oregon
  - Jackson Urological Associates, Jackson, Tennessee
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided